CLINICAL TRIAL: NCT03913260
Title: A Safety, Tolerability, and Pharmacokinetic Study of Different Solution Formulations of LY3375880 Using Investigational Injection Devices in Healthy Subjects
Brief Title: A Study of Different Injectable Formulations of LY3375880 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 17212; I9N-MC-FCAC (Other: Eli Lilly and Company)
Record Dates: First submitted 2019-04-11; First posted 2019-04-12 (Actual); Last update posted 2019-10-11 (Actual); Status verified 2019-10

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: Part A is a crossover design. Part B is a parallel design.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (7):
- Part A: LY3375880 Formulation A (Experimental): LY3375880 Formulation A administered subcutaneously (SC).
  Interventions: Drug: LY3375880; Device: Autoinjector (AI)
- Part A: LY3375880 Formulation B (Experimental): LY3375880 Formulation B administered subcutaneously SC.
  Interventions: Drug: LY3375880; Device: Autoinjector (AI)
- Part A: LY3375880 Formulation C (Experimental): LY3375880 Formulation C administered SC.
  Interventions: Drug: LY3375880; Device: Autoinjector (AI)
- Part A: Positive Control (Placebo Comparator): Positive Control (buffer matrix, only) administered SC.
  Interventions: Drug: Buffer Matrix (No LY3375880); Device: Autoinjector (AI)
- Part B: LY3375880 Test 1 (Experimental): LY3375880 Test 1 Formulation administered SC.
  Interventions: Drug: LY3375880; Device: Manual Syringe
- Part B: LY3375880 Test 2 (Experimental): LY3375880 Test 2 Formulation administered SC.
  Interventions: Drug: LY3375880; Device: Manual Syringe
- Part B: LY3375880 Test 3 (Experimental): LY3375880 Test 3 Formulation administered SC.
  Interventions: Drug: LY3375880; Device: Manual Syringe

INTERVENTIONS:
Drug: LY3375880 — Administered SC
  Arms: Part A: LY3375880 Formulation A; Part A: LY3375880 Formulation B; Part A: LY3375880 Formulation C; Part B: LY3375880 Test 1; Part B: LY3375880 Test 2; Part B: LY3375880 Test 3
Drug: Buffer Matrix (No LY3375880) — Administered SC
  Arms: Part A: Positive Control
Device: Autoinjector (AI) — AI used to administer LY3375880 or Buffer Matrix
  Arms: Part A: LY3375880 Formulation A; Part A: LY3375880 Formulation B; Part A: LY3375880 Formulation C; Part A: Positive Control
Device: Manual Syringe — Manual syringe used to inject LY3375880
  Arms: Part B: LY3375880 Test 1; Part B: LY3375880 Test 2; Part B: LY3375880 Test 3

SUMMARY:
The main purposes of this study are: 1. To learn more about the safety and side effects of different formulations of LY3375880 and 2. To measure how much LY3375880 gets into the blood stream and how long it takes to get out of the body. The study will last about 85 days. Screening may occur up to 28 days prior to enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Are overtly healthy males or females, as determined by medical history and physical examination
* Have a body mass index of 18.0 to 32.0 kilograms per meter squared (kg/m²) inclusive
* Females who are not of child-bearing potential
* Males who agree to use a reliable method of birth control during the study and for 120 days following the final administration of LY3375880
* Are reliable and willing to make themselves available for the duration of the study and are willing to follow study procedures

Exclusion Criteria:

* Have known allergies to LY3375880, related compounds or any components of the formulation, or history of significant atopy
* Have participated or are currently enrolled in clinical trials with LY3375880
* Have infections or evidence of infections
* Are pregnant, lactating or breast feeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-09-19 (Actual); Study Completion 2019-09-19 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) Pain Score | Part A: Within 1-minute post injection
  The pain VAS is a participant administered single item scale designed to measure pain using a 0-100 millimeter (mm) horizontal VAS. Overall severity of participant's pain is indicated by placing a single mark on the scale from 0 mm (no pain) to 100 mm (severe pain).
Pharmacokinetics (PK): Maximum Concentration (Cmax) of LY3375880 | Part B: Predose through Day 85
  PK: Cmax of LY3375880
PK: Area Under the Concentration Versus Time Curve (AUC) of LY3375880 | Part B: Predose through Day 85
  PK: AUC of LY3375880

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (2):
- United States (2):
  - Covance Clinical Research Inc, Daytona Beach, Florida
  - Covance, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No